CLINICAL TRIAL: NCT00127751
Title: A Cardiovascular Disease Multifactor Risk Reduction Program for Medically Underserved High-Risk Patients
Brief Title: Heart Disease on the Mend
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Stanford University (Other)
Collaborators: The Health Trust of Santa Clara County (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 373765
Record Dates: First submitted 2005-08-05; First posted 2005-08-08 (Estimated); Last update posted 2005-08-25 (Estimated); Status verified 2005-08

CONDITIONS: Coronary Heart Disease; Stroke; Hyperlipidemia; Hypertension
Keywords: Risk factor reduction; cardiovascular disease prevention
MeSH Terms: conditions — Coronary Disease; Stroke; Hyperlipidemias; Hypertension

INTERVENTIONS:
Behavioral: Enhance health lifestyle changes and medication compliance

SUMMARY:
The primary objective of this study was to evaluate the effectiveness of a multifactor cardiovascular disease (CVD) risk reduction program using team case management in high risk patients who have low family incomes and limited access to medical care. Patients were randomized to case management (99) or usual care (49) with baseline, 6-month and 12-month evaluations of CVD risk factors, clinical status and quality of life.

DETAILED DESCRIPTION:
The primary objective of this study was to evaluate the effectiveness of a multifactor cardiovascular disease (CVD) risk reduction program using team case management in high risk patients who have low family incomes and limited access to medical care. Patients were randomized to case management (99) or usual care (49) with baseline, 6-month and 12-month evaluations of CVD risk factors, clinical status and quality of life. Subjects were primarily recruited from patients being seen in free medical clinics in Santa Clara County California. Primary eligibility was ≥ 35 years of age, one or more CVD risk factors (with or without clinical CVD), low family income, and residing in Santa Clara County. Patients in the case management group were provided counseling services by specially trained registered nurses (RNs) and registered dieticians (RDs) and assisted in obtaining medications and medical services from programs provided in the county or indigent drug programs provided by selected pharmaceutical companies. Protocol driven treatment algorithms based on national practice guidelines were used and use of existing programs and resources were maximized. On average patients in case management were seen by staff 6-9 in the 12 months.

ELIGIBILITY:
Inclusion Criteria:

* Men and women ≥ 35 years
* One or more major risk factors
* Live in Santa Clara County
* Low family income that limits access to medical care

Exclusion Criteria:

* Under active medical treatment for cancer, CVD or other major medical disorder
* Reasonable access to health care
* Under 35 years of age
* Not a resident of Santa Clara County

Min Age: 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150
Dates: Start 2000-05; Study Completion 2003-05

PRIMARY OUTCOMES:
Cardiovascular disease risk score
Low-density lipoprotein (LDL)-cholesterol
Systolic blood pressure

SECONDARY OUTCOMES:
Body mass index (BMI)
Physical activity score
Nutrition score

CONTACTS AND LOCATIONS:
Overall Officials: William L Haskell, PhD, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States